CLINICAL TRIAL: NCT00372359
Title: Adverse Effect of Prolonged Methylphenidate Treatment on Cardiac Functions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ornit Cohen (Other)
Responsible Party: Sponsor-Investigator, Ornit Cohen, r&d unit, Barzilai Medical Center
Organization: Barzilai Medical Center (Other)
Other Study IDs: BAR1400CTIL
Record Dates: First submitted 2006-09-03; First posted 2006-09-06 (Estimated); Last update posted 2012-09-20 (Estimated); Status verified 2012-09

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Attention Deficit Disorder; Attention Deficit Hyperactivity Disorder; Attention Deficit Disorders With Hyperactivity; Attention Deficit Hyperactivity Disorders
Keywords: Attention Deficit Disorder; Hyperactivity; Methylphenidate
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Spasm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to find out whether prolonged treatment with methylphenidate has any adverse effect on cardiac functions and measurements.

DETAILED DESCRIPTION:
Attention deficit hyperactivity disorder (ADHD) is the most common neurobehavioral condition of childhood, with symptoms consisting of inattentiveness, impulsivity and hyperactivity. The diagnosis relies on subjective criteria since there is no objective test for ADHD. Stimulants are the recommended treatment, during the last 2 decades both the rate of its use has increased, and the age for starting treatment has decreased. Adverse side effects have been few, none of which were serious.

Recently, regulators of the Food and Drug Administration (FDA) have been told on forty deaths among patients who took stimulants through 2003. Accordingly, a subcommittee of the FDA recommended that prescription drugs to treat ADHD should be accompanied by strong 'black-box' warnings that they may increase the risk of heart problems in some patients.

To date, there does not appear to have been any study that has evaluated cardiac functions in these patients. In this study we will evaluate the possible long term effect of methylphenidate on cardiac functions, as to provide more knowledgeable basis for decisions on the treatment of ADHD patients with methylphenidate.

Children age 8-18 years who were treated on methylphenidate for more then five years will be allocated in outpatient clinics. Complete EKG and echocardiographic examinations will be performed and cardiac functions, left ventricular mass and left ventricular muscle width will be compared to the normal range of values. The results will give us, for the first time, a basis to support or reject the causative relationship between these drugs and severe cardiac problems.

ELIGIBILITY:
Inclusion Criteria:

Children with ADHD aged 8-18 years who are taking methylphenydate (Ritalin©, Ritalin SR©, Ritalin LA©) for more than 5 years.

Exclusion Criteria:

Children with any known heart disease or anomaly. Children whose ADHD is part of a syndrome or are mentally retarded. Children that are on any other chronic medications.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged 8-18 that are at least 5 years on methylphenidates
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2006-08; Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Shraga Aviner, MD, PhD, Principal Investigator — The Barzilai Medical Center, Ashkelon, Israel
Locations (1):
- Pediatric Day Care Center, The Barzilai Medical Center, Ashkelon, Israel

REFERENCES:
- [Background] Cohen AL, Jhung MA, Budnitz DS. Stimulant medications and attention deficit-hyperactivity disorder. N Engl J Med. 2006 May 25;354(21):2294-5. doi: 10.1056/NEJMc060860. No abstract available. PMID 16723627
- [Background] Wooltorton E. Medications for attention deficit hyperactivity disorder: cardiovascular concerns. CMAJ. 2006 Jul 4;175(1):29. doi: 10.1503/cmaj.060718. Epub 2006 Jun 13. No abstract available. PMID 16772535
- [Background] Nissen SE. ADHD drugs and cardiovascular risk. N Engl J Med. 2006 Apr 6;354(14):1445-8. doi: 10.1056/NEJMp068049. Epub 2006 Mar 20. No abstract available. PMID 16549404
- [Background] Debate over warnings for ADHD stimulants. Child Health Alert. 2006 Apr;24:1. No abstract available. PMID 16673500